CLINICAL TRIAL: NCT00214305
Title: Effects of Swallowing Therapy in Head and Neck Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-373
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Range of Motion Therapy Program (Experimental): The program involves exercises and maneuvers that include voluntary maximal movements of the tongue, pitch range exercises, head lifting (Shaker exercise), resistance to laryngeal excursion (Mendelsohn Maneuver), breath holding after swallow and cough, thermal-tactile stimulation (ice), suck-swallow, optimal posturing, and dietary changes.
  Interventions: Behavioral: Range of Motion Therapy Program
- Postural Sensory Therapy Program (Placebo Comparator): The program involves all of the above, except that range of motion exercises (voluntary maximal movements of the tongue, pitch range exercises, head lifting, resistance to laryngeal excursion, breath holding after swallow and cough) are not performed.
  Interventions: Behavioral: Postural Sensory Therapy Program

INTERVENTIONS:
Behavioral: Range of Motion Therapy Program — The program involves exercises and maneuvers that include voluntary maximal movements of the tongue, pitch range exercises, head lifting (Shaker exercise), resistance to laryngeal excursion (Mendelsohn Maneuver), breath holding after swallow and cough, thermal-tactile stimulation (ice), suck-swallow, optimal posturing, and dietary changes.
  Arms: Range of Motion Therapy Program
Behavioral: Postural Sensory Therapy Program — The program involves all of the above, except that range of motion exercises (voluntary maximal movements of the tongue, pitch range exercises, head lifting, resistance to laryngeal excursion, breath holding after swallow and cough) are not performed.
  Arms: Postural Sensory Therapy Program

SUMMARY:
Treatment for head and neck cancer often results in significant swallowing problems because of reduced range of motion (ROM) of the larynx, tongue base, and pharyngeal walls. Our question is: Is swallowing therapy to improve ROM during swallowing maneuvers efficacious in patients with reduced ROM?

DETAILED DESCRIPTION:
Patients with head and neck cancer who are treated with chemoradiation and/or surgical resection may exhibit a variety of swallowing difficulties due to reduced range of motion (ROM) resulting from absence or alteration of the structures involved in deglutition. Chemoradiation protocols have been receiving increased attention in the treatment of head and neck cancer. The primary focus of these regimens is disease control and organ sparing. Preservation of oropharyngeal anatomy, however, has not equated with preservation of function. Due to the severity and frequency of swallowing problems in this population, it is critical that the effectiveness of dysphagia (i.e. swallowing disorder) rehabilitation protocols on preservation and/or restoration of function be determined. In the absence of potential remediation, patients may reject organ preservation treatment protocols because of negative functional side effects. There have been a number of therapeutic exercises designed to improve swallowing that have been shown to have a positive effect on head and neck cancer patients who are dysphagic as a result of treatment with surgery and/or chemoradiation. The short- and long-term effectiveness of these exercises has not been defined. The purpose of this study is to compare the effectiveness of combined ROM and postural sensory therapy for swallowing dysfunction to postural sensory therapy alone. By maximizing the effectiveness of therapy, it is expected that improved swallowing function will translate into better quality of life through enjoyment of meals and improved nutrition and hydration so critical to the health and sense of well being of individuals recovering from head and neck cancer.

To be included, subjects must be between 21 and 80 years old and have undergone treatment for the head and neck cancer in the form of chemoradiation, and/or one of the following specific types of head and neck cancer surgery: supraglottic laryngectomy, anterior resection with primary or skin graft closure, anterior resection with distal or free flap closure, posterior resection with primary or skin graft closure, or posterior resection with distal or free flap. Potential subjects must have been diagnosed with Stage I-IV disease and also be available for twice-weekly swallowing therapy sessions. Furthermore, subjects must be available for 12 months while on study.

No subject will be included who has any history of other medical problems that may affect swallowing, speech, voice, neurological problems, gastroenterological problems, or other health problems as determined by the patient's physician and the investigators. Patients with prior treated cancer of the head and neck, or who received a total laryngectomy operation are also not eligible.

ELIGIBILITY:
Inclusion Criteria:

* Subject have undergone treatment for the head and neck cancer in the form of chemoradiation, and/or one of the following specific types of head and neck cancer surgery: supraglottic laryngectomy, anterior resection with primary or skin graft closure, anterior resection with distal or free flap closure, posterior resection with primary or skin graft closure, or posterior resection with distal or free flap
* Potential subjects must have been diagnosed with Stage I-IV disease

Exclusion Criteria:

* history of medical problems that may affect swallowing, speech, voice
* neurological problems
* gastroenterological problems
* prior treatment for cancer of the head and neck
* patient who received a total laryngectomy

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-08

PRIMARY OUTCOMES:
improved swallowing function | 1-month, 4-month, 6-month, and 12-month post treatment

SECONDARY OUTCOMES:
significantly more oral intake | 1-month, 4-month, 6-month, and 12-month post treatment
a less restricted diet | 1-month, 4-month, 6-month, and 12-month post treatment
less cost for medically needed services | 1-month, 4-month, 6-month, and 12-month post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Diane Bless, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States